CLINICAL TRIAL: NCT05923619
Title: Comparison of Post-operative Pain After Total Pulpotomy and Root Canal Treatment in Mature Molars According to New and Traditional Classification of Pulpitis: A Randomized Controlled Trial
Brief Title: Evaluation of Post-operative Pain After Total Pulpotomy and Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Merve Sari, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2308
Record Dates: First submitted 2023-06-16; First posted 2023-06-28 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Post-operative Pain; Pulpitis - Irreversible
Keywords: irreversibl pulpitis; mineral trioxide aggregate; post-operative pain; total pulpotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total pulpotomy (Experimental): The coronal pulp tissue was completely removed with a high-speed sterile carbide bur under abundant water coolant. A cotton pellet moistened with 2.5% sodium hypochlorite was used to achieve hemostasis. Following the achievement of hemostasis, an average of 3 mm thick MTA material (Angelus, Londrina, PR, Brazil) was used to cover the pulp chamber. In the same session, the pulp chamber was closed with approximately 2 mm thick flowable glass ionomer cement (Glass Liner, WP), and coronal restoration was completed with composite filling (Estelıte® Sıgma Quıck, Tokuyama).
  Interventions: Procedure: Total pulpotomy
- Root canal treatment (Active Comparator): The working length was determined using a 15 K type file and apex locator (Morita Root ZX, Tokyo, Japan) and checked by radiography. The chemomechanical preparation was completed using the R25 (Resiproc, VDW, Munich, Germany) file in the mesial root canals and the R25, R40, and R50 files in the distal root canals, respectively, at the WL. During the chemomechanical preparation, the root canals were irrigated with 2.5% NaOCl after every three pecking motions; and total volume of NaOCl was 10 ml. In the final irrigation, the root canal was irrigated with 5 ml 17% Ethylene diamine tetraacetic acid (EDTA), for 1 minute, following with 2 ml distilled water. Following the retention of 5 ml of 2.5% NaOCl in the root canal for 1 minute, 5 ml of distilled used to neutralize the effect of NaOCl in the root canal.Tthe root canals were filled with the lateral condensation using epoxy-resin-based sealer (AH Plus, Dentsply DeTrey GmbH, Konstanz, Germany).
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Total pulpotomy — Total pulpotomy procedures explained in arm descriptions.
  Arms: Total pulpotomy
Procedure: Root canal treatment — Root canal treatment procedures explained in arm descriptions.
  Arms: Root canal treatment

SUMMARY:
The aim of this study was to compare post-operative pain following total pulpotomy (TP) and root canal treatment (RCT) in mature molar teeth with severe symptoms indicative of irreversible pulpitis. To compare the traditional pulpitis classification with the Wolters system in evaluating post-operative pain.

Materials and Methods: Sixty-four mature mandibular molar with symptomatic vital pulps in patients aged 18-60 years were included and were classified according to the Wolters (moderate/severe pulpitis) and the traditional pulpitis classification (reversible/irreversible pulpitis). The teeth randomly divided into 2 groups. RCT was performed, using standardized protocols. TP was performed to the level of the canal orifices, and haemostasis was achieved with 2.5% NaOCl. 3 mm layer of MTA was placed as the pulpotomy agent. The treated teeth were restored with glass ionomer cement followed by composite. Pain was recorded 6, 12, 24, 48, 72 hours and 7 days after treatment. The data collected were statistically analyzed

DETAILED DESCRIPTION:
The literature does not contain any studies comparing the effects of TP and RCT procedures on post-operative pain in mature molar teeth diagnosed with irreversible pulpitis and severe symptoms. Therefore, this study evaluated the effect of pre-operative and intra-operative variables and the treatment method on post-operative pain.

Patient evaluation and treatment procedure

As a result of clinical and radiographic examination, the teeth were classified both according to American Association of Endodontists (AAE) and as proposed by Wolters. The presence/absence of percussion was noted. Pre-operative pain levels were determined according to the Heft-Parker Visual Analog Scale (HP VAS), which consisted of a 10 mm long horizontal line where numerical values were divided into visual categories. Patients were instructed to score their pain with a value on the HP VAS. The presence or absence of pain was classified according to 4 categories:

No pain (level 1, 0), Mild pain (level 2, 1-3 mm), Moderate pain (level 3, 4-6mm), Severe pain (level 4, 7-10 mm). After inferior alveolar nerve block anesthesia was performed with local anesthetic (adrenaline 4% Articaine, 1:100,000), the tooth was isolated with a rubber dam. The isolated area was cleaned using a cotton pellet wetted first with 3% hydrogen peroxide and then 2% chlorhexidine. The entire caries was removed non-selectively using a high-speed diamond bur under water coolant followed by a sterile round steel bur in a slow handpiece. After the pulp exposure was clinically confirmed, the patient was assigned to the TP or RCT group. Randomization was performed using online software with a four-block size block randomization technique to ensure even distribution between the groups (www.randomizer.org). The clinician could not be blinded due to the stages of treatment.

Both patients were prescribed 400 mg of ibuprofen following treatment and asked to use it if necessary. They were informed to consult the clinic in case of severe post-operative pain that was not relieved by analgesics. All participants were administered a questionnaire form based on HP VAS, which could show their pain and analgesic intake after 6 hours, 12 hours, 24 hours, 48 hours, 72 hours, and seven days. Patients were asked to fill in the form. Patients were invited for clinical examination one week after treatment, and follow-up appointments were scheduled for three months, six months, and one year for patients who were observed to be asymptomatic.

ELIGIBILITY:
Inclusion Criteria:

* Standard periodontal pocket depth and mobility,
* Deep/extreme deep caries (periapical radiography),
* Diagnosed with moderate and severe pulpitis according to the Wolters classification,
* Had a positive response to the cold test,
* Mandibular first and second molar teeth with completed root development.

Exclusion Criteria:

* Patients who had received antibiotic therapy in the last three months or used non-steroidal anti-inflammatory drugs within the last twelve hours,
* Patients with diabetes or immunosuppressive disease or pregnancy,
* Teeth that cannot be restored or require post-core,
* Sinus tract or abscess,
* Did not respond to pulp sensitivity test (cold test),
* Teeth with no exposed pulp after non-selective caries removal.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
post-operative pain | 1 week
  Pre-operative and post-operative pain scores were determined according to the Heft-Parker Visual Analog Scale (HP VAS), which consisted of a 10 mm long horizontal line where numerical values were divided into visual categories. Patients were instructed to score their pain with a value on the HP VAS. The presence or absence of pain was classified according to 4 categories:
  No pain (level 1, 0), Mild pain (level 2, 1-3 mm), Moderate pain (level 3, 4-6mm), Severe pain (level 4, 7-10 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Merve Sarı, DDS, Principal Investigator — Department of Endodontics, Faculty of Dentistry, Hatay Mustafa Kemal University; Koray Yılmaz, Study Director — Department of Endodontics, Faculty of Dentistry, Hatay Mustafa Kemal University
Locations (1):
- Department of Endodontics, Faculty of Dentistry, Hatay Mustafa Kemal University, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sabeti M, Huang Y, Chung YJ, Azarpazhooh A. Prognosis of Vital Pulp Therapy on Permanent Dentition: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Endod. 2021 Nov;47(11):1683-1695. doi: 10.1016/j.joen.2021.08.008. Epub 2021 Sep 1. PMID 34478787
- [Background] Levin LG, Law AS, Holland GR, Abbott PV, Roda RS. Identify and define all diagnostic terms for pulpal health and disease states. J Endod. 2009 Dec;35(12):1645-57. doi: 10.1016/j.joen.2009.09.032. PMID 19932339
- [Background] Ricucci D, Russo J, Rutberg M, Burleson JA, Spangberg LS. A prospective cohort study of endodontic treatments of 1,369 root canals: results after 5 years. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Dec;112(6):825-42. doi: 10.1016/j.tripleo.2011.08.003. PMID 22099859
- [Background] Taha NA, Al-Rawash MH, Imran ZA. Outcome of full pulpotomy in mature permanent molars using 3 calcium silicate-based materials: A parallel, double blind, randomized controlled trial. Int Endod J. 2022 May;55(5):416-429. doi: 10.1111/iej.13707. Epub 2022 Mar 17. PMID 35152464
- [Background] Careddu R, Duncan HF. A prospective clinical study investigating the effectiveness of partial pulpotomy after relating preoperative symptoms to a new and established classification of pulpitis. Int Endod J. 2021 Dec;54(12):2156-2172. doi: 10.1111/iej.13629. Epub 2021 Sep 26. PMID 34490637
- [Background] Wolters WJ, Duncan HF, Tomson PL, Karim IE, McKenna G, Dorri M, Stangvaltaite L, van der Sluis LWM. Minimally invasive endodontics: a new diagnostic system for assessing pulpitis and subsequent treatment needs. Int Endod J. 2017 Sep;50(9):825-829. doi: 10.1111/iej.12793. No abstract available. PMID 28776717
- [Background] Parirokh M, Torabinejad M, Dummer PMH. Mineral trioxide aggregate and other bioactive endodontic cements: an updated overview - part I: vital pulp therapy. Int Endod J. 2018 Feb;51(2):177-205. doi: 10.1111/iej.12841. Epub 2017 Sep 21. PMID 28836288
- [Background] Ramani A, Sangwan P, Tewari S, Duhan J, Mittal S, Kumar V. Comparative evaluation of complete and partial pulpotomy in mature permanent teeth with symptomatic irreversible pulpitis: A randomized clinical trial. Int Endod J. 2022 May;55(5):430-440. doi: 10.1111/iej.13714. Epub 2022 Mar 10. PMID 35226769
- [Background] Galani M, Tewari S, Sangwan P, Mittal S, Kumar V, Duhan J. Comparative Evaluation of Postoperative Pain and Success Rate after Pulpotomy and Root Canal Treatment in Cariously Exposed Mature Permanent Molars: A Randomized Controlled Trial. J Endod. 2017 Dec;43(12):1953-1962. doi: 10.1016/j.joen.2017.08.007. Epub 2017 Oct 20. PMID 29061359
- [Derived] Sari M, Yilmaz K, Ozyurek T. Postoperative pain after total pulpotomy and root canal treatment in mature molars according to the new and traditional classifications of pulpitis: a prospective, randomized controlled trial. BMC Oral Health. 2024 Sep 12;24(1):1075. doi: 10.1186/s12903-024-04836-z. PMID 39266985